CLINICAL TRIAL: NCT05799326
Title: Safety and Efficacy of Levofloxacin for Acute Ischemic Stroke: A Randomized Controlled Clinical Trial
Brief Title: Safety and Efficacy of Levofloxacin for Acute Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LVX-AIS
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Levofloxacin
MeSH Terms: conditions — Ischemic Stroke | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levofloxacin group (Experimental): Levofloxacin 200mg twice per day is administrated.
  Interventions: Drug: Levofloxacin
- Levofloxacin simulant group (Placebo Comparator): Levofloxacin simulant 200mg twice per day is administrated.
  Interventions: Drug: Levofloxacin simulant

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin is a quinolone antibiotics and newly identified neuro-protective agent.
  Arms: Levofloxacin group
Drug: Levofloxacin simulant — Levofloxacin simulant is placebo.
  Arms: Levofloxacin simulant group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of levofloxacin in treating acute ischemic stroke.

DETAILED DESCRIPTION:
Acute ischemic stroke is a leading cause of disability and mortality. The investigators' previous studies suggested levofloxacin to be a newly identified neuro-protective agent, which could reduce infarct volume and improve neurologic function in animal models. To evaluate the efficacy and safety of levofloxacin in treating acute ischemic stroke patients, the prospective, multicenter and randomized controlled trial was designed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. The patients were clinically diagnosed with acute ischemic stroke with NIHSS score ≥5 points and ≤15 points,and NHISS score 1a level of consciousness < 1 point.
3. mRS≤1 before stroke onset.
4. Signed and dated informed consent is obtained.

Exclusion Criteria:

1. Patients with transient ischemic attack and those undergoing emergency reperfusion therapy, including intravenous thrombolysis and emergency thrombectomy.
2. Patients using glucocorticoids, antiarrhythmic drugs (class I and class III antiarrhythmic drugs: quinidine, procaine amine, lidocaine, phenytoin sodium, verapamil, etc.), and quinolones within 14 days.
3. Patients with other diseases that may aggravate adverse drug reactions, such as ventricular arrhythmias, prolonged QT interval (male: QTc>430ms, female: QTc>450ms), severe cardiac insufficiency (NYHA functional grade ≥ III), myasthenia gravis, peripheral neuropathy, seizures, tendon-related diseases, severe immune system-related diseases, hematological diseases, active hepatitis or cirrhosis, serious respiratory diseases.
4. Abnormal liver and kidney function: glutamic oxaloacetic transaminase or glutamic pyruvic transaminase exceeds 3 times the upper limit of normal; Direct bilirubin or indirect bilirubin more than 3 times the normal upper limit; Blood creatinine exceeds 1.1 times the upper limit of normal; Creatinine clearance rate≤50ml/min; Urea nitrogen≥ 20mg/dL.
5. Concurrent infection.
6. Blood glucose lower than 3.9 mmol/L.
7. Patients allergy to fluoroquinolones or other antibiotics.
8. Patients with a life expectancy less than 3 months or patients unable to complete the study for other reasons.
9. Not willing to be followed up or poor treatment compliance.
10. Patients who are participating in other clinical studies, or have participated in other clinical studies within 3 months before enrollment, or have participated in this study.
11. Other conditions not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
NIHSS at discharge/7 days | discharge/7 days
  National Institute of Health stroke scale (NIHSS) ranged from 0 to 42, a low value represents a better outcome.

SECONDARY OUTCOMES:
Infarct volume after 3 days of Levofloxacin/simulant treatment | immediately after 3 days of Levofloxacin/simulant treatment
  assessed by magnetic resonance imaging brain scan
Modified rankin scale (mRS) score at 30 days | 30 days
  Modified Rankin Scale (mRS), ranged from 0 to 6, a low value represents a better outcome.
mRS score at 90 days | 90 days
  Modified Rankin Scale (mRS), ranged from 0 to 6, a low value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, PhD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China